1

4

5

6

7 8

9

10

11

12

13

14

15

16

17

18

19

20

21 22

23

24

25

26

27 28

29

30 31

32

## **Research and HIPAA Research Authorization** Supporting Black breast cancer survivors: Feasibility trial of **Study Title:** health coaching-based navigation at the conclusion of treatment

The Ohio State University Combined Consent to Participate in

**Principal Investigator:** Bridget Oppong, MD

Department of Surgery - Division of Surgical Oncology **Sponsor:** 

- This is a consent form for research participation. It contains important information about this study and what to expect if you decide to participate. Please consider the information carefully. Feel free to discuss the study with your friends and family and to ask questions before making your decision whether or not to participate.
- Your participation is voluntary. You may refuse to participate in this study. If you decide to take part in the study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your usual benefits. Your decision will not affect your future relationship with The Ohio State University. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.
- You may or may not benefit as a result of participating in this study. Also, as explained below, your participation may result in unintended or harmful effects for you that may be minor or may be serious depending on the nature of the research.
- You will be provided with any new information that develops during the study that may affect your decision whether or not to continue to participate. If you decide to participate, you will be asked to sign this form and will receive a copy of the form. You are being asked to consider participating in this study for the reasons explained below.

## **Key Information About This Study**

The purpose of this research is to understand the needs and challenges experienced by Black breast cancer survivors through assessing completion of scheduled referrals and participation in support services such as wellness/health coaching. The study navigator will contact you within 48 hours of consent. The wellness/health coach will ask you survey questions about your quality of life, along with questions about how you are doing since your cancer treatment. The interview will last no longer than 60 minutes. After the initial call, the wellness/health coach will reach out with bi-weekly 30-minute coaching sessions for 3 months. Then, monthly sessions for an additional 3 months. Finally, there will be a post-study survey.

#### 1. Why is this study being done?

Black/ African American women experience a 40% higher breast cancer specific mortality compared to white counterparts. Although disparities persist in outcome, breast cancer patients overall continue to benefit from advances in treatment to make breast cancer a survivable disease for most women. The increase in survival combined with the growth and aging of the US population have produced a rise in the number of cancer survivors estimated to be more than 3.8 million women. As the numbers of survivors increase, there are reported unmet supportive care needs, including psychological distress and deficits in physical functioning. To address these needs, many cancer centers offer group coaching and counseling sessions on a variety of topics including psychological services, exercise counseling, and nutrition counseling. While there are limited studies exploring the specific needs of Black breast cancer survivors, the few that exist report a lack of culturally appropriate cancer resources necessary to understand and cope with their diagnosis. We want to evaluate the impact on health coaching on addressing the needs and challenges experienced by Black breast cancer survivors through assessing completion of scheduled referrals and participation in support services.

#### 2. How many people will take part in this study?

We anticipate 40 Black women based on the number of self-identified African American women who present consultation per year.

## 3. What will happen if I take part in this study?

#### Screening & Enrollment

All study procedures are designed to work around your needs and be as flexible as possible in order to best fit into your lifestyle. Breast cancer patients seen in the NP run survivorship clinic will be recruited and consented. The study navigator will contact the participant within 48 hours. A needs assessment will be performed. Based on the needs assessment and the recommendations/ referrals for supportive services from the survivorship NP (formal psychooncology visit or programming of the James Care for Life offerings), the navigator will facilitate scheduling, and outline an individualized plan for the patient.

#### Follow-up

You will be contacted by the wellness/health coach from The Ohio State University over the telephone to complete additional needs, including physical complaints will be addressed by the survivorship clinic providers (NPs) if beyond the scope or comfort of the navigator/coach. "Check in" will be performed with biweekly virtual (30 min) sessions for 3 months and will reduce to monthly sessions until the 6-month period. After the final check-in, you will receive a post-study survey.

# 4. How long will I be in the study?

Your participation in this research study is expected to last for 6-months. This time period will start once you consent to enroll in the study, participate in baseline interview questions and will include telephone follow-up assessments with your health coach. There will be a final, post study survey as well.

## 5. Can I stop being in the study?

 You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University. If you plan to withdraw from the study, please contact **Dr. Bridget Oppong at bridget.oppong@osumc.edu.** 

## 6. What risks, side effects or discomforts can I expect from being in the study?

One risk to you from participating in this study is that private health information about you will be recorded by our study team. We must protect the privacy of health information about you. Health information includes all information about you that is collected during this study. This includes interview responses, medical records and other data that our study team collects. We may use or share your health information for research only if you let us.

Breach of confidentiality is a risk to being in the study if it happens that your information is taken by, given to, or seen by someone who should not be able to look at it or have it. We take all necessary precautions to prevent this, as described in the "Other Information" section below.

Other risks include feeling upset by some of the questions we ask, and being inconvenienced due to the time involved. The research associate or the study investigators will always be available during the study to discuss with you any distress you are experiencing. There is also a risk that you may find the interviews inconvenient. All efforts will be made to make the interviews as easy and short as possible. Our study staff is available in the evenings and on the weekends to complete the telephone interviews if that works best for your schedule.

# 7. What benefits can I expect from being in the study?

The information we gain from this research may help us provide better support to Black breast cancer survivors where the participant can receive additional support in

survivorship in addition to the standard program. There is evidence that interview participants may experience benefits from talking to someone about their perspectives, such as improved self-understanding, a sense of helping others, or feeling they are contributing to science. It is possible that you may not receive any individual benefit from participation in this study.

127 128 129

123

124125

126

#### 8. What other choices do I have if I do not take part in the study?

130131

You may choose not to participate without penalty or loss of benefits to which you are otherwise entitled.

132133134

## 9. What are the costs of taking part in this study?

135136

There is no cost for participating in this study.

137138

#### 10. Will I get paid for taking part in this study?

The team will not remunerate participants for their time. The team anticipates that participants will not incur any expenses during this study.

141

139

140

#### 11. What happens if I am injured because I took part in this study?

142143144

145

If you suffer an injury from participating in this study, you should notify the researcher or study doctor immediately, who will determine if you should obtain medical treatment at The Ohio State University Wexner Medical Center.

146147148

The cost for this treatment will be billed to you or your medical or hospital insurance. The Ohio State University has no funds set aside for the payment of health care expenses for this study.

150151152

149

# 12. What are my rights if I take part in this study?

153154

155

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By signing this form, you do not give up any personal legal rights you may have as a participant in this study.

156157158

159

You will be provided with any new information that develops during the course of the research that may affect your decision whether or not to continue participation in the study.

160161162

You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled.

An Institutional Review Board responsible for human subjects research at The Ohio State University reviewed this research project and found it to be acceptable, according to applicable state and federal regulations and University policies designed to protect the rights and welfare of research participants.

168169170

165

166167

## 13. Will my de-identified information be used or shared for future research?

171172

Yes, it/they may be used or shared with other researchers without your additional informed consent.

173174175

## 14. Will my study-related information be kept confidential?

176177

178179

Efforts will be made to keep your study-related information confidential. However, there may be circumstances where this information must be released. For example, personal information regarding your participation in this study may be disclosed if required by state law.

180 181 182

Also, your records may be reviewed by the following groups (as applicable to the research):

183 184

185

187

• Office for Human Research Protections or other federal, state, or international regulatory agencies;

186

U.S. Food and Drug Administration;
The Ohio State University Institutional Review Board or Office of Responsible Research Practices;

188 189

The sponsor supporting the study, their agents or study monitors; and
Your insurance company (if charges are billed to insurance).

190 191

Tour insurance company (if charges are office to insurance).

192

# 15. HIPAA AUTHORIZATION TO USE AND DISCLOSE INFORMATION FOR RESEARCH PURPOSES

193 194 195

# I. What information may be used and given to others?

196 197

• Past and present medical records;

198

• Research records;

199 200 Records about phone calls made as part of this research;Records about your study visits;

201202

• Information that includes personal identifiers, such as your name, or a number associated with you as an individual;

203

• Information gathered for this research about:

204205

Laboratory, x-ray, and other test results Questionnaires

206

Diagnosis and surgical procedures

207 208

# II. Who may use and give out information about you?

| 2 | 0 | 9 |
|---|---|---|
| 2 | 1 | 0 |

Researchers and study staff.

211212

## III. Who might get this information?

213214

215

216

217

218

219

220

221

222

- The sponsor of this research. "Sponsor" means any persons or companies that are:
  - working for or with the sponsor; or
  - owned by the sponsor.
- Authorized Ohio State University staff not involved in the study may be aware that you are participating in a research study and have access to your information;
- If this study is related to your medical care, your study-related information may be placed in your permanent hospital, clinic, or physician's office record;
- Others: [include specific names of the sponsor, collaborators, study monitor (CRO, SMO), healthcare providers, persons or organizations that analyze health information for the study, data safety monitoring boards, etc..].

223224225

## **IV.** Your information <u>may</u> be given to:

226227

228

229

230

231

232

233

- The U.S. Food and Drug Administration (FDA), Department of Health and Human Services (DHHS) agencies, and other federal and state entities;
- Governmental agencies in other countries;
- Governmental agencies to whom certain diseases (reportable diseases) must be reported; and
- The Ohio State University units involved in managing and approving the research study including the Office of Research and the Office of Responsible Research Practices.

234235236

#### V. Why will this information be used and/or given to others?

237238

239

- To do the research;
- To study the results; and
- To make sure that the research was done right.

240241242

# VI. When will my permission end?

243244245

There is no date at which your permission ends. Your information will be used indefinitely. This is because the information used and created during the study may be analyzed for many years, and it is not possible to know when this will be complete.

246247248

# VII. May I withdraw or revoke (cancel) my permission?

249250

251

Yes. Your authorization will be good for the time indicated above unless you change your mind and revoke it in writing. You may withdraw or take away your permission to use and

disclose your health information at any time. You do this by sending written notice to the researchers. If you withdraw your permission, you will not be able to stay in this study. When you withdraw your permission, no new health information identifying you will be gathered after that date. Information that has already been gathered may still be used and given to others.

256257258

252

253254

255

# VIII. What if I decide not to give permission to use and give out my health information?

259260261

262

Then you will not be able to be in this research study and receive research-related treatment. However, if you are being treated as a patient here, you will still be able to receive care.

263264265

## IX. Is my health information protected after it has been given to others?

266267

There is a risk that your information will be given to others without your permission. Any information that is shared may no longer be protected by federal privacy rules.

268269270

#### X. May I review or copy my information?

271272

Signing this authorization also means that you may not be able to see or copy your study-related information until the study is completed.

274275

273

# 16. Who can answer my questions about the study?

276277278

For questions, concerns, or complaints about the study, or if you feel you have been harmed because of study participation, you may contact **Dr. Bridget Oppong at 614-293-6408.** 

280281282

283

284

279

For questions related to your privacy rights under HIPAA or related to this research authorization, please contact HIPAA Privacy Officer in the College of Medicine Office of Health Sciences, Suite E2140, 600 Ackerman Road, Columbus, Ohio 43202 or by phone at 614-293-4477.

285286287

For questions about your rights as a participant in this study or to discuss other study-related concerns or complaints with someone who is not part of the research team, you may contact the Office of Responsible Research Practices at 1-800-678-6251.

289290291

| and I am aware that I am being ask ortunity to ask questions and have a participate in this study. form. I will be given a copy of this ion form. | had ther |
|---|---|
| | G. |
| | 5 |
| Signature of participant | |
| Date and time | AN |
| Signature of person authorized to consent for (when applicable) | r participar |
| Date and time | AN |
| Simulation of many shadowing and the same of the same | _ |
| Signature of person obtaining consent | |
| Signature of person obtaining consent Date and time | |
| Date and time | AN |
| Date and time I by the IRB | AN |
| Date and time I by the IRB Signature of witness | AN |
| | Signature of person authorized to consent fo (when applicable) |